CLINICAL TRIAL: NCT01060098
Title: T Cells and TNF: The Impact of TNF Blockade on Effector T Cell Populations in Rheumatoid Arthritis and Other Conditions Treated With Anti-TNFalpha Agents
Brief Title: T Cells and TNF (Tumor Necrosis Factor): The Impact of TNF Blockade
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 2104091
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic | interventions — Etanercept; Adalimumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rheumatoid arthritis: Participants with Rheumatoid arthritis
  Interventions: Drug: anti-TNF therapy (etanercept or adalimumab)
- Ankylosing spondylitis: Participants with Ankylosing spondylitis
  Interventions: Drug: anti-TNF therapy (etanercept or adalimumab)
- Psoriatic arthritis: Participants with Psoriatic arthritis
  Interventions: Drug: anti-TNF therapy (etanercept or adalimumab)

INTERVENTIONS:
Drug: anti-TNF therapy (etanercept or adalimumab) — Biological DMARD
  Other Names: Enbrel; Humira

SUMMARY:
We aim to translate these findings into patients with rheumatoid arthritis and other conditions treated with anti-TNF (anti-tumor necrosis factor) therapy, such as psoriatic arthritis and ankylosing spondylitis. Patients from rheumatology clinics within NHS (National Health Service) trusts will be recruited. We will correlate disease activity assessed by clinical parameters, ultrasonography, and questionnaires with biomarkers in the blood and target tissues, such as synovium and skin.

DETAILED DESCRIPTION:
Inflammatory arthritis particularly rheumatoid arthritis (RA), psoriatic arthritis and ankylosing spondylitis are potentially disabling conditions which cause joint pain, swelling and deformity and treatments are aimed at preventing these complications. Although treatment has improved with the advent of anti TNF alpha therapies, up to 30% of patients fail to respond to this treatment and in others, treatment is associated with significant side effects. The precise mechanisms of this remain unclear. In addition, there are no sensitive methods available to monitor or predict disease response to treatment aside from testing inflammatory markers in the blood. Understanding the mechanism of action and what governs response to anti TNF therapy will allow development of more specific therapies for inflammatory arthritis. Work in animal models of rheumatoid arthritis has characterised a novel cell type, Th17 cells, important in the inflammatory cascade which are affected in a particular way by anti TNF therapies and may underpin their mechanism of action and side effects.

ELIGIBILITY:
Inclusion criteria:

* Only anti-TNF naïve patients will be included in this study
* Patients between 18 to 80 years of age
* Patients due to start treatment with anti-TNF blocking agents - etanercept or adalimumab

Patients with rheumatoid arthritis

* Only patients meeting the 1987 American College of Rheumatology (ACR) revised classification criteria for rheumatoid arthritis will be included
* Patients should have active rheumatoid arthritis, defined by an initial DAS28 score >5.1
* Patients should have at least 1 joint suitable for synovial biopsy
* Patients can be on concurrent DMARDs but they should have been on a stable dose of DMARD for at least 1 month prior to study entry
* Patients can be on a concurrent dose of glucocorticoids (up to 10mg daily) and they should have been on a stable dose for at least 4 weeks prior to study entry

Patients with psoriatic arthritis

* Patients should have a secure diagnosis of psoriatic arthritis determined by a rheumatologist
* Patients with psoriatic arthritis included in this study should have evidence of concurrent psoriatic skin lesions at the time of study entry
* Patients should have at least one joint suitable for synovial biopsy
* Patients can be on concurrent DMARDs - they should be on a stable dose of DMARD for at least 1 month prior to study entry

Patients with Ankylosing spondylitis

* Patient should fulfil the Modified New York Criteria for diagnosis of ankylosing spondylitis
* Patients can be on concurrent NSAIDs
* Patients can be on concurrent DMARDs - they should be on a stable dose of DMARD for at least 1 month prior to study entry

Exclusion Criteria:

* Patients who have been previously treated with anti-TNF therapy for whatever reason
* Patients with rheumatoid arthritis, psoriatic arthritis or ankylosing spondylitis who do not fulfil the diagnostic criteria for these conditions as above
* Patient who have received an intra-articular injection of steroids or have received an intra-muscular injection of depot steroid to treat disease flare in the preceding 4 weeks prior to commencing anti-TNF therapy.
* Patients with intercurrent, active infection of any type, excluding the common cold

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Abraham, Principal Investigator — Imperial College London
Locations (1):
- Kennedy Institute Clinical Trials Unit, 4Wl, Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hull DN, Cooksley H, Chokshi S, Williams RO, Abraham S, Taylor PC. Increase in circulating Th17 cells during anti-TNF therapy is associated with ultrasonographic improvement of synovitis in rheumatoid arthritis. Arthritis Res Ther. 2016 Dec 23;18(1):303. doi: 10.1186/s13075-016-1197-5. PMID 28010726
- [Result] Hull DN, Williams RO, Pathan E, Alzabin S, Abraham S, Taylor PC. Anti-tumour necrosis factor treatment increases circulating T helper type 17 cells similarly in different types of inflammatory arthritis. Clin Exp Immunol. 2015 Sep;181(3):401-6. doi: 10.1111/cei.12626. Epub 2015 Jun 23. PMID 25766640

RESULTS

PARTICIPANT FLOW:
Groups:
- Rheumatoid Arthritis: Participants with Rheumatoid arthritis anti-TNF therapy (etanercept or adalimumab): Biological DMARD
Period: Overall Study
Arm/Group | Rheumatoid Arthritis | Ankylosing Spondylitis | Psoriatic Arthritis
Started | 25 | 15 | 8
Completed | 25 | 15 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthritis | Ankylosing Spondylitis | Psoriatic Arthritis | Total
Number analyzed (Participants) | 25 | 15 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (11.7) | 36.4 (11.8) | 50.9 (8.4) | 48.23 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 3 | 5 | 26
  Male | 7 | 12 | 3 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25 | 15 | 8 | 48

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Effector T Helper Type 17 Cells in Peripheral Blood
Description: The frequency of circulating Th17 cells was determined by IL17 enzyme-linked immunospot assay (Elispot) and flow cytometry (fluorescence-activated cell sorting (FACS)).
Time Frame: Week 0, Week 12
Population: Patients with RA were studied at protocol visits during the initial 12 weeks of anti-TNF treatment
Measure: Mean (Standard Error); unit: spSFC/10^6
Arm/Group | Rheumatoid Arthritis | Ankylosing Spondylitis | Psoriatic Arthritis
Number analyzed (Participants) | 25 | 15 | 8
spSFC/10^6
  Week 0 | 466.4 (277.6) | 432 (474) | 450 (276)
  Week 12 | 759.8 (510) | 651 (532) | 609 (373)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis; week 0 compared to week 12; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Ankylosing Spondylitis; week 0 compared to week 12; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Psoriatic Arthritis; week 0 compared to week 12; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Rheumatoid Arthritis | Ankylosing Spondylitis | Psoriatic Arthritis
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/15 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/15 | 0/8
Other Adverse Events (participants affected / at risk) | 0/25 | 0/15 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes